CLINICAL TRIAL: NCT04276753
Title: A Randomized, Double-blinded, Placebo Controlled, Monocentric Study to Evaluate the Anti-ageing and Skin Brightening Benefit of the Test Product in Healthy Female Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ratan K. Chaudhuri (Industry)
Responsible Party: Sponsor-Investigator, Ratan K. Chaudhuri, Director, Sytheon Ltd.
Organization: Sytheon Ltd. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: SKIN/SYAS/2020-01
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Skin Aging
MeSH Terms: interventions — chebulae fruit

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terminalia Chebula fruit extract (Experimental): The test product is an emulsion. It contains Terminalia Chebula fruit extract.
  Test product will be applied topically on full face twice a day for 8 weeks.
  Interventions: Other: Terminalia Chebula Fruit Extract
- Placebo (Placebo Comparator): The placebo product is an emulsion with same appearance as the experimental product but without Terminalia Chebula fruit extract.
  Placebo emulsion will be applied topically on full face twice a day for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Terminalia Chebula Fruit Extract — Standardized fruit extract
  Arms: Terminalia Chebula fruit extract
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Every day the cells of the outer layer of skin die off, shed, and regenerate. When young, skin cells turn over quickly, but that turnover rate begins to slow with age, beginning as early as twenties. As a result, skin loses its luster and begins to look dull. Aging caused by the genes is inherited and is called intrinsic (internal) aging. The other type of aging is known as extrinsic (external) aging and is caused by environmental factors, such as exposure to the sun's rays.

Skin ageing is mainly characterized by -

1. Decrease in thickness, firmness & elasticity of skin which results in wrinkles.
2. Reduction in antioxidant capacities.
3. Formation of spider veins and dark circles under the eyes. This study is proposed to evaluate skin antiaging efficacy along with the brightening attributes on face by visual assessment by Dermatologist, image analysis using VISIA CR, skin elasticity by Cutometer (MPA580) Hydration by Corneometer and skin texture by Antera 3 D and skin lightening/fairness by spectrophotometer, water barrier function by TEWL and to skin pH level by pH meter.

DETAILED DESCRIPTION:
Every day the cells of the outer layer of skin die off, shed, and regenerate. When young, skin cells turn over quickly, but that turnover rate begins to slow with age, beginning as early as twenties. As a result, skin loses its luster and begins to look dull. Aging caused by the genes is inherited and is called intrinsic (internal) aging. The other type of aging is known as extrinsic (external) aging and is caused by environmental factors, such as exposure to the sun's rays.

Skin ageing is mainly characterized by -

1. Decrease in thickness, firmness & elasticity of skin which results in wrinkles.
2. Reduction in antioxidant capacities.
3. Formation of spider veins and dark circles under the eyes.

The epidermis, dermis and subcutaneous tissues are the top, middle and bottom layers of the skin respectively. The top layer shows the wrinkles, age spots, deep lines, and depressions. The skin dermis contains macromolecules, polysaccharides, glycosaminoglycans (GAGs), fibrous protein (collagens, elastin), salts and water which together are known as the extra cellular matrix, responsible for tissue cohesion.

The subcutaneous tissues contain fatty deposits. Another part of the skin is the sebaceous glands that produce sebum which lubricates the skin and keeps it soft and smooth. All three skin layers contribute to the aging process. As a person gets older, less sebum is produced, and this makes the epidermis drier. Dry skin is more prone to wrinkling.

Signs of ageing include facial wrinkles, pigmentation, fine lines, crow's feet and Nasolabial folds. Ageing also impacts texture and elasticity of the skin.

Skin lightening or skin brightening, refer to the application of topical products in an attempt to lighten skin tone and provide an even skin complexion by reduction in melanin. The glow is not dependent on the skin colour of the person, i.e. a darker skin tone person can have very good Skin Glow. However, pigmentation errors like uneven skin tone, blemishes, blotchiness and spots also results in varied reflectance of light from the skin surface and results in dullness of the skin. It is also known that skin hydration, skin texture and pigmentation concerns can impact the skin glow. This study is based on evaluating Skin glow based on the relationship of these attributes.

This study is proposed to evaluate skin antiaging efficacy along with the brightening attributes on face by visual assessment by Dermatologist, image analysis using VISIA CR, skin elasticity by Cutometer (MPA580) Hydration by Corneometer and skin texture by Antera 3 D and skin lightening/fairness by spectrophotometer, water barrier function by TEWL and to skin pH level by pH meter.

ELIGIBILITY:
Inclusion Criteria:

* Female adult subjects in general good health as determined from a recent medical history, general physical examination, dermatological assessment.
* Subjects in the age group of 35-50 years (both ages inclusive).
* Subject with Fitzpatrick skin types III to V (ITA to be recorded at forehead and flexor forearm)
* Subjects with chronic pollution exposure in past 5 years based on pollution questionnaire (Refer annexure 1)
* Subjects with normal to dry skin type (corneometer reading upto 35)
* Subjects with mild to moderate fine lines and wrinkles in periorbital area (Crow's feet-under eye) & forehead (Refer annexure 3 for photonumerical scale)
* Subjects with minimum one spot with width ≥3 mm
* Subjects with chronic pollution exposure in past 5 years based on pollution questionnaire (Refer annexure 1)
* Subject free of excessive hair, acne, cuts, abrasions, fissures, wounds, lacerations, or any other active skin conditions on the face.
* Subject who agrees not to use any other product/treatment/home remedy/ except the provided product on their face during the study period other than the test product.
* Subjects who agree not to carry out bleaching or any other procedures including facial etc. on face during the study period.
* Subjects who agree not to expose to excessive sun light. (Sun exposure not more than half an hour daily and during that time use of umbrella to cover face).
* Subjects willing to give a voluntary written informed consent, photography release and agree to come for regular follow-up.
* Subjects willing to abide by and comply with the study protocol.

Exclusion Criteria:

* Subject with any other signs of significant local irritation or skin disease.
* Subject currently taking any medication, which the Investigator believes may influence the interpretation of the data.
* Subject having clinically significant systemic or cutaneous disease, chronic illness or had major surgery in the last year.
* Subjects who do not agree to remove all jewellery on/around face (e.g., necklace, earrings, if possible nose ring), during VISIA imaging.
* Subjects having hair style which covers almost the entire forehead
* Subjects undergoing any treatment of any skin condition on their face/forearm.
* Subjects not willing to discontinue other topical facial products.
* Subject allergic or sensitive to bar cleansing products, cosmetics, creams/lotions, artificial jewellery or anything else.
* Pregnant women (as confirmed by UPT) and lactating women
* Subjects on any medical treatment either systemic/topical in the past 1 month or currently taking medication including food supplements.
* Subjects with skin allergy history or atopic dermatitis or psoriasis
* Subjects who have participated in any other clinical trial in the last 3 months.
* Subjects using oral contraceptive pills or hormonal implants as birth control measures during the study
* Subjects that was treated with Botox/filler /bio stimulatory molecules injection

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 26 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the investigational product for skin aging benefits | 8 weeks
  Evaluate the antiaging effect of investigational product in 8 weeks w.r.t baseline in comparison to placebo as per below parameters.
  i. Skin texture ii. Signs of aging iii. Skin elasticity/Firmness iv. Skin wrinkles and expression lines v. Skin dryness
Evaluate the investigational product for skin brightening benefits | 8 weeks
  Evaluate the skin brightening benefit of investigational product in 8 weeks w.r.t. baseline in comparison to placebo as per below parameters.
  i. Glow and radiance ii. Evenness iii. Clarity iv. Skin colour

SECONDARY OUTCOMES:
Evaluate the product safety and tolerance by skin tolerance evaluation by dermatologist. | 8 weeks
  Evaluate the product safety and tolerance by skin tolerance evaluation by dermatologist.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mukesh Ramnane, MD, Principal Investigator — MSCR
Locations (1):
- MSCR, Bengaluru, Karnatka, India

IPD SHARING:
Plan to Share IPD: No